CLINICAL TRIAL: NCT05665127
Title: Point of Care Evaluation of High-sensitivity Cardiac Troponin
Acronym: POC-ET
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); NHS Grampian (Other Government); Siemens Healthcare Diagnostics Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: AC21114; RG/20/10/34966 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2022-12-06; First posted 2022-12-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this observational research project the investigators wish to test new technologies that could allow them to either detect or rule out heart attacks earlier.

Currently, when a patient attends the Emergency Department with symptoms that could be due to a heart attack, the patient has a blood test taken from a vein in the arm. This is sent to a laboratory to measure the level of a protein called troponin that is released from the heart when it is damaged. Doctors and nurses use the level of troponin measured in that blood sample, along with a tracing of the heart and an assessment of symptoms, to decide whether the patient is having a heart attack. On average, it takes about 2 hours from the patient arriving at hospital to the doctor or nurse receiving the blood test result so they can make this diagnosis.

A device has been designed that can measure troponin by using a drop of blood from a finger prick with the result available in around 10 minutes. This means that if a patient is having a heart attack we can diagnose it earlier and give them treatment. Previous studies have also showed that the majority of patients who attend hospital with chest pain ultimately do not have a heart attack. With this new device the investigators hope to be able to reassure these patients that their symptoms are not due to a heart attack, so the clinical team can concentrate on finding out what else could be causing their chest pain, and ultimately discharge them earlier.

The investigators aim to find the best way to use this new device and look at the impact this device has on the length of time from sample to diagnosis and time spent in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to hospital with symptoms of suspected acute coronary syndrome
* Age 18 years and over

Exclusion Criteria:

* Patients with ST-segment elevation on the electrocardiogram
* Patients presenting with an out-of-hospital cardiac arrest
* Patients unable or unwilling to give informed consent
* Patients unable or unwilling to comply with study protocol
* Previous enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected acute coronary syndrome attending the Emergency Department or Acute Medical Unit
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Type 1, 4b or 4c myocardial infarction or cardiac death | Index presentation to 30 days

SECONDARY OUTCOMES:
Any myocardial infarction | Index presentation to 1 year
Cardiac death | Index presentation to 1 year
Any myocardial infarction or cardiac death | Index presentation to 1 year
Cardiovascular death | Index presentation to 1 year
All-cause death | Index presentation to 1 year
Reattendance with suspected acute coronary syndrome | Index presentation to 1 year
Unplanned coronary revascularization | Following index presentation to 1 year

OTHER OUTCOMES:
Time from presentation to rule-out or rule-in myocardial infarction | Time of index presentation until the time of reporting of the troponin result that rules in or rules out myocardial infarction, assessed up to the end of study follow up (12 months)
Duration of stay in hospital (index) | Time from index presentation until the time of discharge from hospital, assessed up to the end of study follow up (12 months)
Duration of stay in Emergency Department | Time from index presentation until the time of discharge from the Emergency Department, assessed up to the end of study follow up (12 months)
Inter-assay coefficient of variation | During index admission, assessed up to 36 hours following enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mills, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No